CLINICAL TRIAL: NCT03024489
Title: A Phase I/II Dose Escalation Study of the CDK4/6 Inhibitor, Palbociclib in Combination With Cetuximab and Intensity Modulated Radiation Therapy (IMRT) for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Palbociclib With Cetuximab and IMRT for Locally Advanced Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA2016001
Record Dates: First submitted 2016-11-28; First posted 2017-01-18 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer; Locally Advanced
Keywords: Phase I/II
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — palbociclib; Cetuximab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Palbociclib-Cetuximab-IMRT (Experimental): * IMRT will be administered 5 days on/2 days off with a total dose of 70 Gy for 33-35 fractions.
  * Cetuximab will be administered 400 mg/m2 IV at 7 days before (day -7) starting radiation and then 250 mg/m2 IV weekly for 7 weeks.
  * Palbociclib will be administered orally daily 3 week-on and 1-week of during IMRT (Day 1-21 and Day 29-49) on 3 dose levels and the MTD.
  Interventions: Drug: Palbociclib; Drug: Cetuximab; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: Palbociclib — Dose Level -1: 100 mg oral every other day 3 week-on and 1-week of during IMRT (Day 1-21 and Day 29-49).
  Other Names: PD-0332991
Drug: Palbociclib — Dose Level 1: 75 mg per oral daily 3 week-on and 1-week of during IMRT (Day 1-21 and Day 29-49).
  Other Names: PD-0332991
Drug: Palbociclib — Dose Level 2: 100 mg per oral daily 3 week-on and 1-week of during IMRT (Day 1-21 and Day 29-49).
  Other Names: PD-0332991
Drug: Palbociclib — Dose Level 3: 125 mg per oral daily 3 week-on and 1-week of during IMRT (Day 1-21 and Day 29-49).
  Other Names: PD-0332991
Drug: Cetuximab — All dose levels: 400 mg/m2 IV at 7 days before (day -7) starting radiation and then 250 mg/m2 IV weekly for 7 weeks.
  Other Names: Erbitux
Radiation: Intensity Modulated Radiation Therapy — 5 days on/2 days off with a total dose of 70 Gy for 33-35 fractions.
  Other Names: IMRT

SUMMARY:
Cyclin D kinase 4 (CDK4) is a key regulator of the G1-S transition in the cell cycle. Alterations in CDK4-cyclin D-retinoblastoma (Rb) pathway may lead to carcinogenesis in many cancers. Several mechanisms have been described: (i) Amplification or overexpression of cyclin D1, (ii) Amplification of CDK4, (iii) Activating mutation of CDK4, and (iv) Loss of the CDK4 inhibitor, p16 (CDKN2A). Human Papilloma Virus (HPV) plays a major role in squamous cell carcinoma of head and neck (SCCHN) carcinogenesis. It induces many alterations in the CDK4-Cyclin D-Rb and apoptotic pathways such as up-regulation of p16, loss of Rb and p53 functions. A novel therapy for HPV-negative SCCHN is clearly an unmet medical need.

Palbociclib (PD 0332991) is an orally active, highly selective inhibitor of the CDK4/6 with ability to block Rb phosphorylation in the low nanomolar range. The most advanced development is in a treatment of metastatic breast cancer. In addition, palbociclib showed a radiosensitization property. Since combination of cetuximab and radiation improved PFS and overall survival (OS) in locally advanced SCCHN when compared with radiation alone, these provide a strong rationale to evaluate a combination of palbociclib, cetuximab, and radiation for locally advanced SCCHN. Because many genetic alterations in SCCHN significantly involve in the CDK4-cyclin D-Rb pathway, predictive biomarker(s) of palbociclib in this combination will be explored.

Thus, the investigators propose a non-randomized, dose escalation, phase I study designed to determine the maximum tolerated dose (MTD) and toxicity of palbociclib, cetuximab, and IMRT for locally advanced SCCHN.

DETAILED DESCRIPTION:
The enrollment of an initial patient cohort of 3 or 6 patients will follow the traditional "3 + 3" dose escalation scheme (see table below). The patients will be treated with palbociclib, cetuximab, and IMRT at starting at Dose Level (DL) 1. Subsequent patient cohort(s) will be enrolled depending on the safety and tolerability of the initial cohort. If <33% patients treated at Dose Level 1 experience DLT (see definition below) by the end of treatment (56 days), then next cohort of 3 patients will be enrolled and treated at Dose Level 2. If 2 treatment-related DLTs are observed at Dose Level 1, patients will be accrued to Dose Level -1. The MTD is defined as the maximum dose level at which ≤1/6 patients have DLTs.

At the MTD or RP2D, we will accrue up to 15 locally advanced unresectable p16-negative SCCHN patients to allow for definitive evaluation of tolerability, correlative endpoints and preliminary efficacy. CT/PET scan will be performed at 3 months after the last dose of radiation to evaluate residual disease. Patients with residual disease will be considered for salvage surgery following standard of care.

* IMRT will be administered 5 days on/2 days off with a total dose of 70 Gy for 33-35 fractions.
* Cetuximab will be administered 400 mg/m2 IV at 7 days before (day -7) starting radiation and then 250 mg/m2 IV weekly for 7 weeks.
* Palbociclib will be administered orally daily 3 week-on and 1-week of during IMRT (Day 1-21 and Day 29-49).

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced histology or cytology proven squamous cell carcinoma of oral cavity, oropharynx, larynx, and hypopharynx.
2. Locally advanced SCCCH patients who would be considered for concurrent cetuximab and IMRT as a definitive treatment.
3. Age ≥ 18 yeas old.
4. Available tissue to determine HPV status and the other biomarkers of interest.
5. ECOG status ≤ 1.
6. Adequate bone marrow, liver, and renal functions, defined as:

   * Platelet count ≥150 x 109/L, Absolute Neutrophile Count (ANC) ≥1.5 x 109/L, Hgb ≥9 gm/dL
   * ALT and AST ≤ 1.5 upper limit normal (ULN); serum total bilirubin ≤ ULN
   * Serum creatinine ≤ 1.5 x ULN, or calculated or measured creatinine clearance (by Cockcroft-Gault Equation) ≥ 50 mL/min
   * Magnesium ≥ the lower limit of normal
7. Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of study drug.
8. Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 6 months after last investigational drug dose received.
9. Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

Potential subjects who meet ANY of the following exclusion criteria are not eligible for enrollment into this study:

1. SCCHN patients with distance metastasis.
2. Major surgery < 4 weeks or minor surgery < 2 weeks prior to the first day of study treatment.
3. Patients with previous chemotherapy for cancer treatment and radiation to the head and neck areas.
4. Patients who were previously treated with any CDK4/6 inhibitors or cetuximab.
5. SCCHN with expressed p16 by IHC (only in expansion cohort).
6. Active cardiac disease described as:

   * Left ventricular ejection fraction (LVEF) < 50% by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO).
   * QTc > 480 msec on screening EKG (using the QTcF formula).
   * Congenital long QT syndrome
   * Myocardial infarction or active uncontrolled angina pectoris within the last 6 months prior to the first day of study treatment
   * Uncontrolled significant cardiac arrhythmias except for benign premature ventricular contractions (PVC) and premature atrial contractions (PAC).
   * Symptomatic pericarditis
   * History of cardiomyopathy
7. Weight loss more than 10% from baseline body weight before illness.
8. Active clinically serious infections or other serious uncontrolled medical conditions.
9. Substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results.
10. Unable to swallow an intact palbociclib tablet.
11. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of palbociclib.
12. Known HBV, HCV, and/or HIV infection.
13. Patients who are currently treated with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
14. Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pomelos, or exotic citrus fruits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of dose-limiting toxicities (DLTs) and recommended phase II dose (RP2D) | From baseline to the completion of radiotherapy (up to 8 weeks)
  To describe the dose-limiting toxicities and identify the recommended phase I dose (RP2D) of the combination of palbociclib, cetuximab, and IMRT for locally advanced SCCHN.
  Recommended Phase II Dose (RP2D) is a maximum tolerated dose (MTD) or the highest dose level when MTD is not reached.
  Toxicity will be assessed using the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. A DLT is defined by the occurrence of any of the following toxicities related to palbociclib and the combination within 8 weeks of treatment duration.

SECONDARY OUTCOMES:
Evaluate preliminary efficacy of the combination | From baseline to 3 months after completion of radiotherapy (up to 5 months)
  Objective response rate (ORR) by the RECIST criteria version 1.1 and PET/CT scan response at 3 months after completion of treatment will be used to evaluate preliminary efficacy of this combination.
Evaluate safety profile of the combination of palbociclib, cetuximab and IMRT | From baseline to 1 year after completion of radiotherapy (up to 14 months)
  All toxicities, including acute and chronic toxicities will be evaluated by the CTCAE V.4.
Evaluate anti-tumor activity of the combination depending on Rb status | From baseline to 3 months after completion of radiotherapy (up to 5 months)
  Objective response rate (ORR) by the RECIST criteria version 1.1 and PET/CT scan response at 3 months after completion of treatment will be used to evaluate preliminary efficacy of this combination. Rb status will be correlated with the ORR.

CONTACTS AND LOCATIONS:
Overall Officials: Nuttapong Ngamphaiboon, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ngamphaiboon N, Pattaranutaporn P, Lukerak S, Siripoon T, Jinawath A, Arsa L, Shantavasinkul PC, Taonam N, Trachu N, Jinawath N, Kositwattanarerk A, Sananmuang T, Jiarpinitnun C. A Phase I Study of the CDK4/6 Inhibitor Palbociclib in Combination with Cetuximab and Radiotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma. Clin Cancer Res. 2024 Jan 17;30(2):294-303. doi: 10.1158/1078-0432.CCR-23-2303. PMID 37982827